CLINICAL TRIAL: NCT05478798
Title: Comparison of Three Methods of Fetal Weight Estimation in Patients With Severe and Morbid Obesity
Brief Title: Comparison of Three Methods for Fetal Weight Estimation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Inshirah Sgayer, Dr Inshirah Sgayer, Western Galilee Hospital-Nahariya
Other Study IDs: NHR
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Fetal Weight; Obesity, Morbid; Pregnancy Related
Keywords: fetal weight estimation; ultrasound; maternal subjective estimation; term pregnancy; clinical estimation
MeSH Terms: conditions — Fetal Weight; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ultrasonographic fetal weight estimation — An ultrasonographic estimate will be performed in our ultrasound unit and a calculation by the ultrasound machine is based on Hadlock's formula including measurement of biparietal diameter (BPD), head circumference (HC), abdominal circumference (AC) and femur length (FL).
Other: clinical fetal weight estimation — A clinical weight estimate will be performed by using Leopold's maneuvers
Other: maternal subjective fetal weight estimation — the pregnant woman will tell her subjective estimation of fetal weight estimation

SUMMARY:
The aim of this study was to compare maternal, clinical and ultrasound estimations of fetal weight in women with severe (BMI>35) and morbid (BMI>40) obesity and to determine the effect of maternal body mass index (BMI) on these estimations.

DETAILED DESCRIPTION:
Accuracy of fetal weight estimation is of key importance in antenatal care, as well as in the planning and management of labor and mode of delivery. In order to achieve more accurate prenatal fetal weight estimations and align these with a risk-optimizing mode of delivery, additional tools supporting the standard of use with ultrasound are needed.

The main ultrasonic methods used to calculate the weight of a fetus are based on measurement of fetal abdominal circumference (AC) and estimated fetal weight (EFW) using a formula first described by Hadlock, and the sufficient accuracy of this model has recently been proven.

Leopold's maneuvers have a long-standing tradition in obstetrics and midwifery. By placing both hands on the woman's abdomen the examiner can describe the position of the fetus as well as the level of the uterine fundus and thus detect a disproportion between fetus and the female pelvis. Experienced examiners are able to give a clinical estimation of fetal weight after performing Leopold's maneuvers including symphysis-fundal height and abdominal palpation. Maternal body mass index (BMI) has been shown to affect the accuracy of EFW. For example overweight (BMI>25) patients had found an absolute % error >10% in fetal weight estimation in 42.2% and 24.4% of cases, using Leopold's maneuvers and ultrasound, respectively. Maternal estimation of the fetus weight is as accurate as physicians; clinical estimations, and is advised as a complementary method of assessment. The aim of this study was to compare maternal, clinical and ultrasound estimations of fetal weight in women with severe (BMI>35) and morbid (BMI>40) obesity and to determine the effect of maternal body mass index (BMI) on these estimations.

Pregnant women ≥ 37 weeks and with BMI ≥ 35 with singleton who are admitted before delivery will be offered to participate in the study.

1. A clinical weight estimate will be performed by a trained professional physician using Leopold's maneuvers.
2. An ultrasonographic estimate will be performed in our ultrasound unit and a calculation by the ultrasound machine is based on Hadlock's formula [3] including measurement of biparietal diameter (BPD), head circumference (HC), abdominal circumference (AC) and femur length (FL).
3. For maternal estimate, patients will be asked to give a fetal weight estimation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 37 weeks
* BMI ≥ 35
* Singleton pregnancies
* Fetal weight estimate within two weeks from delivery

Exclusion Criteria:

* Primiparity
* Women who will give birth in a different hospital
* Multiple pregnancy
* Moderate to severe polyhydramnios
* Severe fetal malformations - such as hydrocephalus, hydrops fetalis
* Maternal age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women in term singleton pregnancy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
fetal actual birth weight | immediately after delivery
  fetal actual birth in grams

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sgayer I, Francis YN, Ashkar-Majadla N, Tuma R, Lowenstein L, Frank Wolf M, Odeh M. Three Methods of Fetal Weight Estimation Compared in Women With BMI >/= 35 kg/m2 at Term-A Prospective Observational Study. Birth. 2025 Nov 25. doi: 10.1111/birt.70041. Online ahead of print. PMID 41287954